CLINICAL TRIAL: NCT01928550
Title: Pilot Study OCT of Retinal Blood Flow in Proliferative Diabetic Retinopathy Before and After Panretinal Photocoagulation
Brief Title: Diabetes PRP and OCT
Acronym: PRP
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Oregon Clinical and Translational Research Institute (Other)
Responsible Party: Principal Investigator, David Huang, Christina Flaxel, MD, Oregon Health and Science University
Other Study IDs: IRB00009572; 8UL1TR000128-07 (NIH)
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Diabetes; OCT; PDR
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PDR patients: Patients suspected to have Proliferative Diabetic Retinopathy or PDR

SUMMARY:
The purpose of this study is to evaluate the effectiveness of investigational Doppler Optical Coherence Tomography (OCT) and OCT angiography in the management of proliferative diabetic retinopathy (PDR - a leading cause of blindness in diabetic patients) before and after treatment. Angiography is the mapping of the blood vessels, and Doppler detects blood flow. PDR is due to poor oxygen circulation in smaller blood vessels in the back of the eye (retina), and is observed in 80% of people who have had diabetes for more than 10 years. This study will look at how blood flow to the eye is affected before and after treatment.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) refers to changes in the blood vessels of the retina associated with long-term diabetes mellitus. These changes can be found in patients both with Type I and II diabetes. DR is a leading cause of blindness in the United States. It is categorized as either non-proliferative (NPDR) or proliferative (PDR). In the PDR progress, the lack of oxygen in the retina causes fragile, new blood vessels to grow along the retina and in the clear, gel-like vitreous humour. Without timely treatment, the new vessels can bleed, cloud vision, and destroy the retina. So, the PDR is classified as either the existence of retinal neovascularization or vitreous or pre-retinal hemorrhage. PDR is typically treated with a laser, known as panretinal photocoagulation (PRP), which will create 1,600-2,000 burns in the retina to reduce the retinal oxygen demand, and then reduce the possibility of ischemia, or with an injection of an anti-vascular endothelial growth factor (anti-VEGF) drug into the vitreous, which always needs multiple injections. In cases of severe bleeding, a vitrectomy may be performed under local anesthesia. However, an eye patch and medicated eye drops are always needed after the operation to protect against infection and the outcomes are not always as good as expected.

PDR is currently diagnosed by a comprehensive eye exam including a visual acuity test, ophthalmoscopy or fundus photography, fluorescein angiography (FA) and optical coherence tomography (OCT). If the PDR is thought to require treatment, the subsequent assessment of disease severity and treatment planning utilizes FA. FA requires the injection of sodium fluorescein into the systemic circulation. However, 1 in 3 people have adverse reactions to sodium fluorescein, which can include nausea, vomiting, hives, and acute hypotension. Severe reactions such as anaphylaxis and related anaphylactoid reactions, causing cardiac arrest and sudden death due to anaphylactic shock, have also been reported. Finally, because the risks of sodium fluorescein to a developing fetus are unknown, its use in pregnant women is contraindicated. Replacing FA with a less invasive and better tolerated method would reduce the risk in the patient population. One option is OCT angiography.

Optical coherence tomography is an imaging technology that can perform non-contact cross-sectional imaging of tissue structure in real time. It has a number of features that make it attractive as a diagnostic imaging modality: 1) It has micron-level resolution, which is not possible with any other non-contact technique; 2) No potentially allergenic dyes or contrast agents are required; 3) OCT images are generated in electronic form, which facilitates the use of digital image processing techniques to extract quantitative parameters regarding the imaged tissue anatomy. For these reasons, structural OCT is already routinely used to assess the early stage of DR (NPDR) by imaging the areas of macular edema and response to treatment. Novel functional OCT including Doppler OCT and OCT angiography may allow an assessment of retinal blood flow and alleviate the need for the more invasive FA test. Thus, if the diagnostic data provided by functional OCT are at least equivalent or superior to those achieved by FA, patients and healthcare providers could realize a substantial benefit in utilizing this technology in the management of PDR and the evaluation of PRP.

Therefore, we propose a pilot study to evaluate the feasibility of Doppler OCT to measure total retinal blood flow to assess global retinal ischemia after PRP treatment and OCT angiography of the retina to assess proliferative changes in the management of PDR subjects in comparison to standard FA. Functional OCT data (Doppler OCT and OCT angiography) are acquired using the Swept Source-OCT (SS-OCT) with a depth resolution of 5 microns and an ultrafast scan rate of 100 kHz which allows us to obtain detailed 3D OCT images. OCT angiography performs noninvasive microcirculation measurement and visualization which are not options on commercially available OCT systems. Though not FDA-approved, the SS-OCT prototype satisfies the American national standards for laser safety (ANSI) safety requirement. The power level is low enough to be classified as a non-significant risk device.

ELIGIBILITY:
Inclusion Criteria:

a. Diagnosis of diabetes mellitus (type 1 or type 2).

Exclusion Criteria:

1. Inability to give informed consent.
2. Inability to maintain stable fixation for OCT imaging.
3. Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
4. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
5. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, subject can become eligible.
6. Systemic anti-VEGF or pro-VEGF treatment within 4 months prior to treatment
7. Women who are pregnant or lactating or intending to become pregnant within the next 12 months due to unknown safety of fluorescein angiography
8. Subject is expecting to move out of the area of the clinical center to an area and not willing to return for follow-up visits during the 6 months of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals 18 years of age and older presenting to the Retina Service within the Department of Ophthalmology at the Casey Eye Institute of Oregon Health & Science University with signs and symptoms of PDR will be considered and evaluated for enrollment into this study. This pilot study has a planned enrollment target sample size of 28 subjects needing PRP. However, up to 40 subjects will be recruited as it is possible that after subjects sign the consent form they may not meet all eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
Total retinal blood flow & visual acuity | 1 year
  1) Total retinal blood flow, as measured by Doppler OCT, will be correlated with visual acuity and the severity of PDR. This will be performed by the following analysis:
  1. Pearson's correlation test of total retinal blood flow with logMAR (Logarithm of the Minimal Angle of Resolution) visual acuity before and after PRP;
  2. Pearson's correlation test of total retinal blood flow with area of capillary drop-out on FA before and after PRP;
  3. Pearson's correlation test of total retinal blood flow with areas of leakage on FA before and after PRP;
  4. Pearson's correlation test of total retinal blood flow with areas of thickening on OCT before and after PRP.
  5. Paired t test of total retinal blood flow on OCT before and after PRP.

SECONDARY OUTCOMES:
Macular ischemic areas and microaneurysms, as identified by FA vs. OCT | 1 year
  2) Macular ischemia and retinal neovascularization, as measured by OCT angiography, will be correlated with visual acuity and macular ischemia as evaluated by fluorescein angiography. This will be performed by the following analysis:
  1. Pearson's correlation test of retinal neovascularization identified by OCT angiograms with that identified by FA.
  2. Pearson's correlation test of macular ischemic area with area of capillary drop-out on FA before and after PRP.
  3. Pearson's correlation test of retinal parafoveal flow index and size of retinal neovascularization with logMAR visual acuity before and after PRP;
  4. Paired t test of retinal parafoveal flow index before and after PRP.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States